CLINICAL TRIAL: NCT03171753
Title: Anxiety, Preoperative Stress and Music Therapy
Brief Title: Preoperative Anxiety and Music Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Aggregate Professor, PhD, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5/CE/2016
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders | interventions — Pain Measurement; Clinical Laboratory Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music therapy (Experimental): Listening prerecorded music through an individual headset for 30 min in before the induction of anesthesia
  Interventions: Diagnostic Test: questionnaire; Diagnostic Test: laboratory test; Diagnostic Test: cardiac monitoring; Diagnostic Test: skin resistance; Device: Music listening
- Control (Active Comparator): patients wear headphones for 30 minuts without any sound
  Interventions: Diagnostic Test: questionnaire; Diagnostic Test: laboratory test; Diagnostic Test: cardiac monitoring; Diagnostic Test: skin resistance; Device: No sound

INTERVENTIONS:
Diagnostic Test: questionnaire — questionnarie will be performed before the application of headphone and after their removal.
Diagnostic Test: laboratory test — laboratory test will be collected before the application of headphone and after their removal. the cardiac monitoring will be performed during the all study period
Diagnostic Test: cardiac monitoring — the cardiac monitoring will be performed through study period
Diagnostic Test: skin resistance — the skin resistance monitoring will be performed through study period
Device: Music listening — Listening prerecorded music through an individual headset for 30 min
  Arms: Music therapy
Device: No sound — No sound through an individual headset for 30 min
  Arms: Control

SUMMARY:
Music can reduce anxiety in adult patients awaiting surgical interventions. The study was designed to test the difference in cardiac parameters, anxiety questionnaire, laboratory enzymes, skin resitance between surgical patients listening music vs no sound.

DETAILED DESCRIPTION:
Patients undergoing elective surgical intervention will be allocated in two groups: Group M will listen prerecorded music through an individual headset for 30 min before the induction of anesthesia; Group C will listen no sound through an individual headset for 30 min before the induction of anesthesia The degree of stress and anxiety the patients will be assessed using questionnaire. Laboratory enzymes will be measured.

Heart rate, non invasive arterial pressure, pulse oximetry,skin resistance will be recorded. All the patients will receive continuous ECG holter recording .

To assess the effect of music therapy on the degree of autonomic modulation, HRV will be analyzed with traditional time and frequency measures.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients >18 years old, after obtaining informed consent

Exclusion Criteria:

* patients with hearing impairment,
* any known psychiatric or memory disorder
* thyroid disease.
* atrial fibrillation
* pace-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
cardiac monitoring | through study period (to 15 min before the application of headphones until 15 minutes after their removal
  cardiac variability

SECONDARY OUTCOMES:
questionnaire | questionnaire score change 15 min after the removal of headphones from baseline ( early before the application of headphones)
  anxiety questionnarie
laboratory test | enzyme level change early after the application of headphones from baseline (early before the application of headphones)
  enzyme dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti, Foggia, FG, Italy

IPD SHARING:
Plan to Share IPD: Undecided